CLINICAL TRIAL: NCT07059559
Title: Efficacy of Rhythmic Walking Program on Renal Function and Oxidative Stress in Subjects With Chronic Kidney Disease
Brief Title: Rhythmic Walking Program and Renal Function and Oxidative Stress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Burapha University (Other)
Responsible Party: Principal Investigator, Piyapong Prasertsri, Associate Professor Dr., Burapha University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BRO 2024-074
Record Dates: First submitted 2025-07-01; First posted 2025-07-11 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Renal Function

STUDY DESIGN:
Intervention Model Description: This study is a randomized controlled trial. Patients who consent to participate and pass the screening process will be randomly assigned to groups based on the order of their participation (random by sequence). Patients who join in odd-numbered order, such as 1st, 3rd, 5th, etc., will receive standard care as provided by the hospital (control group). Patients who join in even-numbered order, such as 2nd, 4th, 6th, etc., will receive a walking program.
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors were blinded to the intervention administered to each patient.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Patients who join in odd-numbered order, such as 1st, 3rd, 5th, etc., will receive standard care as provided by the hospital (control group).
- Rhythmic walking group (Experimental): Patients who join in even-numbered order, such as 2nd, 4th, 6th, etc., will receive a walking program. This involves continuous walking exercise for 30 minutes, once a day, three days a week, over a period of three months. During the walking sessions, patients will walk at a pace of 60 steps per minute, or one step per second.
  Interventions: Other: Rhythmic walking

INTERVENTIONS:
Other: Rhythmic walking — Patients who consent to participate and pass the screening process were randomly assigned to groups based on the order of their participation (random by sequence): control group or rhythmic walking group.
  Arms: Rhythmic walking group

SUMMARY:
This study designed a over-knee automatic step counter device. Then, we evaluated its efficacy on renal function and oxidative stress in patients with chronic kidney disease.

DETAILED DESCRIPTION:
This study is a randomized controlled trial. Patients who consent to participate and pass the screening process will be randomly assigned to groups based on the order of their participation (random by sequence). Patients who join in odd-numbered order, such as 1st, 3rd, 5th, etc., will receive standard care as provided by the hospital (control group). Patients who join in even-numbered order, such as 2nd, 4th, 6th, etc., will receive a walking program. This involves continuous walking exercise for 30 minutes, once a day, three days a week, over a period of three months. During the walking sessions, patients will walk at a pace of 60 steps per minute, or one step per second.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Aged between 18 and 59 years
* Diagnosed by a physician with chronic kidney disease stage 2-4, with a glomerular filtration rate (GFR) between 15-89 milliliters per minute, persisting for at least 3 months

Exclusion Criteria:

* No musculoskeletal disorders that hinder walking, such as osteoarthritis
* Not engaging in regular exercise (less than 3 times per week or less than 150 minutes per week)
* Not regularly taking medications or supplements containing antioxidants

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2024-07-17 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2025-07-01 (Actual)

PRIMARY OUTCOMES:
Creatinine level | Day 0 and day 91
  Blood creatinine level was measured in mg/dL unit
Malondialdehyde level | Day 0 and day 91
  Blood malondialdehyde level was measured in micromolar unit
Superoxide dismutase activity level | Day 0 and day 91
  Blood superoxide dismutase activity level was measured in percent unit
Estimated glomerular filtration rate level | Day 0 and day 91
  Estimated glomerular filtration rate level was measured in ml/min/1.73 m2 unit
Estimated creatinine clearance level | Day 0 and day 91
  Estimated creatinine clearance level was measured in ml/min unit

CONTACTS AND LOCATIONS:
Overall Officials: Piyapong Prasertsri, Ph.D., Principal Investigator — Faculty of Allied Health Sciences, Burapha University
Locations (1):
- Rehabilitation Medicine Department, Chamni Hospital, Chamni, Changwat Buri Ram, Thailand

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data (IPD) available to other researchers.